CLINICAL TRIAL: NCT03815409
Title: Rehabilitation of Parkinsonian Gait in Body Weight Support Combined With Treadmill: a Controlled Study
Brief Title: Treadmill in the Rehabilitation of Parkinsonian Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treadmill2007
Record Dates: First submitted 2019-01-07; First posted 2019-01-24 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWSTT group (Experimental): The sessions were conducted on a treadmill with partial weight unload.
  Interventions: Other: Treadmill with partial weight unload
- Control group (Other): The traditional PT rehabilitation treatment included passive, active and active-assisted exercises, according to the methods commonly used (Kabat, Bobath).
  Interventions: Other: Traditional PT rehabilitation treatment

INTERVENTIONS:
Other: Treadmill with partial weight unload — 10-minute treadmill walk with a support corresponding to 20% of his/her own weight, followed by a 5-minute rest and a second 10-minute session on the treadmill with a support corresponding to 10% of his/her own weight. In the initial treadmill session, the starting speed of the treadmill was set to 0.5 km/h, subsequent increments of 0.5 km/h per minute were added to reach the maximum speed that was comfortably tolerated by the patient. This latter was used for the entire training period.
  Arms: BWSTT group
Other: Traditional PT rehabilitation treatment — Every 40-minute treatment session consisted in isotonic and isometric exercises for the major muscles of the limbs and trunk including cardiovascular warm-up exercises (5 minutes), muscle stretching exercises (10 minutes), muscle stretching exercises for functional purposes (10 minutes), balance training exercises (10 minutes), relaxation exercises (5 minutes)
  Arms: Control group

SUMMARY:
Gait disorders represent disabling symptoms in Parkinson's Disease (PD). The effectiveness of rehabilitation treatment with Body Weight Support Treadmill Training (BWSTT) has been demonstrated in patients with stroke and spinal cord injuries, but limited data is available in PD. The aim of the study is to investigate the efficacy of BWSTT in the rehabilitation of gait in PD patients. Thirty-six PD inpatients were enrolled and performed rehabilitation treatment for 4 weeks, with daily sessions. Subjects were randomly divided into two groups: both groups underwent daily 40-minute sessions of traditional physiokinesitherapy followed by 20-minute sessions of overground gait training (Control group) or BWSTT (BWSTT group). The efficacy of BWSTT was evaluated with clinical scales and Computerized Gait Analysis (CGA). Patients were tested at baseline (T0) and at the end of the 4-week rehabilitation period (T1).

DETAILED DESCRIPTION:
Gait disorders in Parkinson Disease (PD) are due to dopaminergic nigrostriatal pathways degeneration and represent important components of the disability.

In PD, gait is characterized by a significant reduction of stride length. Inadequate flexion at the ankle and knee, reduction of heel strike, forward-flexed trunk, reduced arm swing with asymmetric stride times for lower limbs and significant stride-to-stride variability are frequently associated.

The efficacy of pharmacological treatment with Levodopa is frequently incomplete and adjuvant rehabilitation treatment is recommended. Body weight-supported treadmill training (BWSTT) represents a promising rehabilitative approach for gait impairment in PD. Effectiveness of BWSTT on gait, balance and motor function has been demonstrated in different neurological diseases, especially in stroke and spinal cord injury. In PD patients, BWSTT has been tested in small controlled studies that have suggested a clinically detectable beneficial effect. BWSTT seems also effective in improving balance in PD. In PD, many data in literature show how treadmill training, acting as a sensory cue, improves kinetic and kinematic parameters, studied with computerized gait analysis (CGA) more than physiotherapy alone.

The first report of BWSTT efficacy in gait rehabilitation of PD belongs to Miyai. Ten patients with PD were enrolled in a cross-over study and treated for 4 consecutive weeks with BWSTT (20% of unweighting for 12 minutes followed by another 12-min period of 10% of unweighting) or conventional physical therapy (CPT). The Authors showed that BWSTT was superior to CPT in improving gait disturbances and disability at the end of the rehabilitative period. More specifically BWSTT proved superior to CPT in improving UPDRS scores, gait speed and stride length. The same study group in 2002 evaluated the 6-month retention of BWSTT in PD. Twenty-four patients with PD were randomized to receive BWSTT (20% of unweighting for 10 minutes + 10% of unweighting for 10 minutes + 0% of unweighting for an additional 10-min period) or CPT 3 times/week for 4 consecutive weeks. All patients were clinically evaluated at baseline and them monthly for 6 months. In this series, gait speed significantly improved in BWSTT respect to CPT only at month 1, while the improvement in the stride length was more marked in BWSTT group with respect to CPT and persisted until month 4.

In 2008 Fisher speculated on the possible central mechanism responsible for clinical effects f BWSTT. Thirty subjects affected by PD were randomly assigned to three groups: high-intensity group (24 sessions of BWSTT), low-intensity group (24 sessions of CPT), zero-intensity group (8 weeks of education classes). Again, the high-intensity group improved the most at the end of treatment period, in particular in gait speed, step length, stride length and double support. Of note, that in this study a subgroup of patients was also tested with transcranial magnetic stimulation: in the BWSTT group Authors were able to record a lengthening of the cortical silent period, postulating that high-intensity training improved neuronal plasticity in PD, through BDNF and GABA modulation.

Ustinova published the first positive case report on the short-term gait rehabilitation efficacy of BWSTT delivered to a PD patient with a robotic device (Lokomat - Hocoma Inc., Volketswil, Switzerland). The intervention consisted in a 2-week gait training, delivered 3 times per week, with each session lasting 90 to 120 minutes.

Lo conducted a pilot study to assess the efficacy of BWSTT delivered with the Lokomat unit in reducing frequency of freezing (FOG) of gait in PD. Authors reported a 20% reduction in the average number of daily episodes of FOG and a 14% improvement in the FOG-questionnaire score.

In 2012 Picelli enrolled 41 PD patients in the first randomised controlled study aimed to compare the efficacy of BWSTT delivered with a robot-assisted gait training (RAGT - gait Trainer GT1) to CPT (not focused on gait training) in improving gait in PD. They showed how RAGT was significantly superior respect to CPT in improving the 6-minute walking test, the 10-meter walking test, stride length, single/double support ratio, Parkinson's Fatigue Scale and UPDRS score.

In the present study subjects were enrolled among consecutive PD patients hospitalized in the Neuro-Rehabilitation Unit of the IRCCS Mondino Foundation of Pavia, Italy. Thirty-six patients affected by Idiopathic PD, according to the UK Brain Bank diagnostic criteria were included. Subjects were randomly assigned to two groups: 18 PD patients were assigned to the "BWSTT group" and 18 patients to the "Control group". Before starting treatment, patients of BWSTT group performed a 20-minute single session of BWSTT in order to test feasibility and tolerability. Four of them did not tolerate BWSTT: one patient reported an increase in his pre-existing hip pain, two patients with pre-existing spondyloarthrosis complained of low back pain, one patient reported that the procedure induced anxious symptoms. These 4 patients were re-allocated to the control group, so that the final disposition of patients in the two groups was as follows: 14 patients (8 women and 6 men) in the BWSTT group and 22 patients (10 women and 12 men) in the Control group.

Patients in both groups underwent 5 daily rehabilitation sessions per week for 4 consecutive weeks. Both groups underwent daily 40-minute sessions of traditional physical therapy (PT) followed by a 20-minute session of overground gait training (Control group) or of gait training with BWSTT (BWSTT group).

The traditional PT rehabilitation treatment included passive, active and active-assisted exercises, according to the methods commonly used (Kabat, Bobath) and previously published (25, 26) Every 40-minute treatment session consisted in isotonic and isometric exercises for the major muscles of the limbs and trunk including cardiovascular warm-up exercises (5 minutes), muscle stretching exercises (10 minutes), muscle stretching exercises for functional purposes (10 minutes), balance training exercises (10 minutes), relaxation exercises (5 minutes). This protocol was designed in accordance with PD rehabilitation guidelines and evidences in the literature.

The sessions were conducted on a treadmill with partial weight unload. Specifically, the patient performed 10-minute treadmill walk with a support corresponding to 20% of his/her own weight, followed by a 5-minute rest and a second 10-minute session on the treadmill with a support corresponding to 10% of his/her own weight. In the initial treadmill session, the starting speed of the treadmill was set to 0.5 km/h, subsequent increments of 0.5 km/h per minute were added to reach the maximum speed that was comfortably tolerated by the patient. This latter was used for the entire training period.

All patients were examined by a neurologist with expertise in Movement Disorders at the beginning of hospitalization (T0) and at the end of the neurorehabilitation period (+4 weeks, T1). The clinical assessment involved a complete neurological examination and administration of the following clinical scales, validated for the assessment of the damage/disability:

* for the assessment of PD severity: the Unified Parkinson's Disease Rating Scale, part III (UPDRS-III);
* for the assessment of functional independence: the Functional Independence Measure (FIM).

The instrumental assessment of gait was conducted at T0 and T1 by an experienced laboratory Technician using an Optokinetic Gait Analysis System associated to the software Myolab Clinic (ELITE, BTS Engineering Milan), composed of six infrared cameras, with a sampling rate of 100 Hz. According to the Davis protocol, twenty-one spherical reflective markers (15mm in diameter) were applied along the body. Synchronized data acquisition and data processing were performed by analyzer software (BTS, Milan, Italy). In order to perform kinematic analysis of gait, patients were instructed to walk at their preferred speed along a 10-meter walkway with the initial step on the side of disease onset. For each session, the investigators acquired at least three performances and calculated the mean. In order to obtain the best individual performance, all recordings were conducted in the ON phase. The sessions were recorded at 5-min intervals to allow complete recovery from fatigue.

ELIGIBILITY:
Inclusion Criteria:

* disease stage 2-3 Hoehn &Yahr in the "on" phase;
* stable dosage of dopaminomimetic drugs for 3 months before study enrollment

Exclusion Criteria:

* moderate to severe cognitive impairment (MMSE ≤ 21),
* advanced PD (Hoehn and Yahr [H&Y] stage >3),
* unpredictable motor fluctuations
* moderate to severe orthopedic problems or other pathological conditions (e.g. severe postural abnormalities) that might affect gait training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11-15 (Actual); Primary Completion 2008-11-30 (Actual); Study Completion 2008-11-30 (Actual)

PRIMARY OUTCOMES:
speed of gait | after 4-week rehabilitative program
  m/s - higher values represent better outcome

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale III (UPDRS-III) | after 4-week rehabilitative program
  Motor disability of Parkinson's Disease (scale from 0 to 56). Higher values represent a worse outcome.
Functional Independence Measure (FIM) | after 4-week rehabilitative program
  Independence in activity of daily living (scale from 18 to 126). Higher values represent a better outcome.
Cadence of step | after 4-week rehabilitative program
  step/min - higher values represent better outcome
stride duration | after 4-week rehabilitative program
  ms - higher values represent worse outcome
stride length | after 4-week rehabilitative program
  meter - higher values represent better outcome
stance | after 4-week rehabilitative program
  percentage variation - higher values represent worse outcome
swing | after 4-week rehabilitative program
  percentage variation - higher values represent better outcome
number of strides in 10 meters | after 4-week rehabilitative program
  number - higher values represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Study Director — IRCCS Mondino Foundation, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris ME. Movement disorders in people with Parkinson disease: a model for physical therapy. Phys Ther. 2000 Jun;80(6):578-97. PMID 10842411
- [Background] Knutsson E, Lindblom U, Martensson A. Lioresal and spasticity. Acta Neurol Scand Suppl. 1972;51:449-50. No abstract available. PMID 4514375
- [Background] Miyai I, Fujimoto Y, Ueda Y, Yamamoto H, Nozaki S, Saito T, Kang J. Treadmill training with body weight support: its effect on Parkinson's disease. Arch Phys Med Rehabil. 2000 Jul;81(7):849-52. doi: 10.1053/apmr.2000.4439. PMID 10895994
- [Background] Ganesan M, Pal PK, Gupta A, Sathyaprabha TN. Treadmill gait training improves baroreflex sensitivity in Parkinson's disease. Clin Auton Res. 2014 Jun;24(3):111-8. doi: 10.1007/s10286-014-0236-z. PMID 24659140
- [Background] McIntosh GC, Brown SH, Rice RR, Thaut MH. Rhythmic auditory-motor facilitation of gait patterns in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 1997 Jan;62(1):22-6. doi: 10.1136/jnnp.62.1.22. PMID 9010395
- [Result] Bowes SG, Clark PK, Leeman AL, O'Neill CJ, Weller C, Nicholson PW, Deshmukh AA, Dobbs SM, Dobbs RJ. Determinants of gait in the elderly parkinsonian on maintenance levodopa/carbidopa therapy. Br J Clin Pharmacol. 1990 Jul;30(1):13-24. doi: 10.1111/j.1365-2125.1990.tb03738.x. PMID 2202385
- [Result] Miyai I, Fujimoto Y, Yamamoto H, Ueda Y, Saito T, Nozaki S, Kang J. Long-term effect of body weight-supported treadmill training in Parkinson's disease: a randomized controlled trial. Arch Phys Med Rehabil. 2002 Oct;83(10):1370-3. doi: 10.1053/apmr.2002.34603. PMID 12370870
- [Result] Toole T, Maitland CG, Warren E, Hubmann MF, Panton L. The effects of loading and unloading treadmill walking on balance, gait, fall risk, and daily function in Parkinsonism. NeuroRehabilitation. 2005;20(4):307-22. PMID 16403997
- [Result] Mehrholz J, Kugler J, Storch A, Pohl M, Hirsch K, Elsner B. Treadmill training for patients with Parkinson's disease. Cochrane Database Syst Rev. 2015 Sep 13;2015(9):CD007830. doi: 10.1002/14651858.CD007830.pub4. PMID 26363646
- [Result] Ganesan M, Sathyaprabha TN, Pal PK, Gupta A. Partial Body Weight-Supported Treadmill Training in Patients With Parkinson Disease: Impact on Gait and Clinical Manifestation. Arch Phys Med Rehabil. 2015 Sep;96(9):1557-65. doi: 10.1016/j.apmr.2015.05.007. Epub 2015 May 23. PMID 26008873
- [Result] Bartolo M, Serrao M, Tassorelli C, Don R, Ranavolo A, Draicchio F, Pacchetti C, Buscone S, Perrotta A, Furnari A, Bramanti P, Padua L, Pierelli F, Sandrini G. Four-week trunk-specific rehabilitation treatment improves lateral trunk flexion in Parkinson's disease. Mov Disord. 2010 Feb 15;25(3):325-31. doi: 10.1002/mds.23007. PMID 20131386
- [Result] Tassorelli C, De Icco R, Alfonsi E, Bartolo M, Serrao M, Avenali M, De Paoli I, Conte C, Pozzi NG, Bramanti P, Nappi G, Sandrini G. Botulinum toxin type A potentiates the effect of neuromotor rehabilitation of Pisa syndrome in Parkinson disease: a placebo controlled study. Parkinsonism Relat Disord. 2014 Nov;20(11):1140-4. doi: 10.1016/j.parkreldis.2014.07.015. Epub 2014 Aug 13. PMID 25175601
- [Derived] Berra E, De Icco R, Avenali M, Dagna C, Cristina S, Pacchetti C, Fresia M, Sandrini G, Tassorelli C. Body Weight Support Combined With Treadmill in the Rehabilitation of Parkinsonian Gait: A Review of Literature and New Data From a Controlled Study. Front Neurol. 2019 Feb 8;9:1066. doi: 10.3389/fneur.2018.01066. eCollection 2018. PMID 30800095